CLINICAL TRIAL: NCT05110508
Title: Active KC: a Text Message Based Intervention for Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jordan Carlson, Study Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001939
Record Dates: First submitted 2021-09-09; First posted 2021-11-08 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Physical Activity; Patient Engagement
Keywords: text message; technology; Garmin; physical activity
MeSH Terms: conditions — Motor Activity; Patient Participation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical Activity Self-Regulation (Experimental): Participants will receive multiple weekly text messages. Texts will contain wear reminders, encouragements, congratulatory content, and behavior change messages based on the Garmin data. Some text message content asks for a response from the participant to help tailor later messages for behavior change support.
  Interventions: Behavioral: Text Based Behavioral Intervention for Physical Activity

INTERVENTIONS:
Behavioral: Text Based Behavioral Intervention for Physical Activity — Text intervention messaging will be sent through an automated text messaging service programmed by the CM Informatics team, which has been approved by the institution. Participants will be asked to wear Garmin physical activity monitor to provide physical activity information throughout the intervention. The Garmin is worn like a wristwatch. The device is small and non-intrusive. The Garmin device is a consumer wearable that will automatically detect and track activity such as walking, running, and cycling. The text messages incorporate information from the Garmin monitor to support physical activity.

SUMMARY:
Active KC will involve delivering PA support tools to individuals interested in increasing their physical activity. The tools involve provision of a Garmin wearable activity monitor and participant-tailored behavior change supports (e.g., goal setting and monitoring) delivered through text messaging and a corresponding study website.

ELIGIBILITY:
Inclusion Criteria:

* Individual has a smart device with internet or data and app downloading and texting capability
* Can read or write in English
* At least 8 years old (there is no upper age limit)
* Willing to complete study measures, participate in intervention, and share data collected in Active KC with the main study

Exclusion Criteria:

* Does not meet the above inclusion criteria
* Non-adherent to study measurement (wearing the Garmin less than 4 days) during baseline period
* Averaging over 60 minutes per day of physical activity (children) or 30 minutes of physical activity per day (adults) during the baseline period as measured by the Garmin
* Participant has a disability that interferes with their ability to carry out daily activities

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in Physical Activity Minutes Over Time | 8 weeks
  Participant physical activity will be measured by daily minutes of physical activity as collected by the Garmin monitor.
Changes in Physical Activity Steps Over Time | 8 weeks
  Participant physical activity will be measured by a daily step count as collected by the Garmin monitor.

SECONDARY OUTCOMES:
Participant Engagement of Text Messages | 8 weeks
  Text message engagement as measured by number of texts responded to.
Views of Participants on Intervention Preferences via Participant Survey | Baseline, End of Study (8 weeks)
  Adults will complete a baseline and follow up adult survey and children will complete a baseline and follow up child survey with help from their caregiver when appropriate. Participant surveys may be distributed via hardcopy, email, or text message.
Participant Engagement of the Garmin Monitor | 8 weeks
  Garmin activity monitor engagement as measured by number of wear days.
Views of Participants on intervention via Focus Groups | Week 4, Week 8
  Up to 15 focus groups will be hosted throughout and after the intervention period. A subsample of participants will be selected to take part in focus groups conducted after week 4 and week 8. These focus groups will ask about participant experiences with the Garmin monitors and text messaging along with general perceptions of the intervention. Focus groups will be hosted virtually using Teams or in person and will be recorded. All participants will have the option to keep their cameras off during virtual focus groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States